CLINICAL TRIAL: NCT07325032
Title: Effectiveness of Deep Breathing and Three Typical Yoga Poses for Kinesiophobia Among Knee Osteoarthritis Patients
Brief Title: Impact of Breathing and Yoga Poses on Kinesiophobia in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Snekha V, Primary investigator, Saveetha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 332/07/2024/ISRB/UGSR/SCPT
Record Dates: First submitted 2025-12-15; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Kinesiophobia; Osteo Arthritis Knee
Keywords: Kinesio phobia; Osteoarthritis; Mind body practice; Yoga poses; Deep breathing technique; Conventional physiotherapy; Physical and emotional stability
MeSH Terms: conditions — Kinesiophobia; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Breathing technique and conventional physiotherapy (Active Comparator): Participants received Deep Breathing exercise and conventional physiotherapy for five times per week for four weeks with rest periods.
  Interventions: Behavioral: Deep Breathing exercise
- Three Yoga poses and conventional physiotherapy (Active Comparator): Participants received Three Typical yoga poses and conventional physiotherapy for five days each, for a total of four weeks with rest periods.
  Interventions: Behavioral: Three typical yoga poses

INTERVENTIONS:
Behavioral: Deep Breathing exercise — The participants are seated on chair were given a 3-min, 6 deep breaths per minute along with the Conventional physiotherapy protocol 5 times a week for 4 weeks.
  Other Names: Conventional physiotherapy
  Arms: Deep Breathing technique and conventional physiotherapy
Behavioral: Three typical yoga poses — The participants were asked to perform three typical yoga poses on yoga mat along with the Conventional physiotherapy protocol 5 times a week for 4 weeks.
  Other Names: Conventional physiotherapy
  Arms: Three Yoga poses and conventional physiotherapy

SUMMARY:
The study aimed to determine if deep breathing and conventional physiotherapy were more effective than yoga poses and conventional physiotherapy in reducing kinesiophobia among knee osteoarthritis patients. 40 participants were divided into an experimental and control group, with the experimental group receiving deep breathing exercise and conventional physiotherapy, and the control group receiving yoga poses and conventional physiotherapy.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative joint disease causing severe pain, stiffness, and functional limitations. It involves synovial proliferation, cartilage degeneration, and structural joint changes. Knee OA is influenced by age, limb use, injury, mechanical stress, genetics, and metabolic factors, with varied clinical presentations. The knee is a complex joint made of the femoropatellar and medial/lateral femorotibial joints. It functions as a condylar synovial joint with tibial and femoral condyles, and also includes menisci that divide the joint space, increasing complexity.

Women are more likely to develop OA, with the knee being the most commonly affected. Around 344 million people require rehabilitation for OA. With rising obesity and injury rates, global OA prevalence is expected to increase. In India, OA rates differ significantly between rural and urban regions. Daily function in OA is affected not only by physical damage but also by psychological factors. Fear and avoidance behaviors can worsen pain, contributing to kinesiophobia and negatively impacting mobility.

Kinesiophobia is an excessive fear of movement or reinjury due to beliefs about pain or harm. It occurs in conditions like shoulder pain, chronic low back pain, and aging. The Tampa Scale for Kinesiophobia (TSK) is used to assess this fear.

Deep breathing relaxation techniques, including slow inhalation, breath-holding for ~5 seconds, and gentle exhalation, help reduce anxiety by relaxing supporting muscles. Deep breathing promotes emotional control, calmness, better metabolism, and regulates pain and mood through autonomic pathways.

Deep, slow breathing (DSB) can reduce pain, improve mood, and enhance sleep in healthy individuals and OA patients. It is cost-effective, calming, and may reduce joint tension, encouraging better participation in physical activity. Yoga, a mind-body practice with roots in India, enhances balance, coordination, mood, strength, flexibility, and range of motion. Pranayama (breathing) and asanas (postures) together improve both physical and mental well-being. It is considered safe for people of all ages.

Physiotherapy and exercise have been used for nearly a century to treat knee osteoarthritis. They are the second most prescribed treatment after medication. However, the long-term effectiveness and benefits of supervised, home-based, or independent exercise remain uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 - 60
* Documented diagnosis of Osteoarthritis
* Tampa scale Score =<68
* Pain severity score 7-10(severity) on Visual Analog Scale
* Short-form McGill Pain Questionnaire (SF-MPQ-2): =<220

Exclusion Criteria:

* Severe Joint Deformity or Instability
* Recent Surgery or Injury
* Severe Range of Motion (ROM) Limitations
* Neurological Conditions
* Cardiovascular or Respiratory Conditions

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Tampa scale for kinesiophobia | Baseline and week 4
  Tampa scale is a 17-item self-reported instrument used to distinguish between non-excessive fear and phobia in patients with chronic musculoskeletal pain, i.e., the fear of movement. Each item is a 4 -point scale anchored from 1 (strongly disagree) to 4 (strongly agree) with total score of 68. The Score 17 and below representing (no kinesiophobia) and for a participants from score 37- 68 (represents kinesiophobia).

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline and week 4
  The Visual Analogue Scale is a widely used tool for measuring pain severity, with endpoints ranging from "no pain" to "worst pain imaginable." Patients mark points on the scale, and clinicians track changes over time.

OTHER OUTCOMES:
Short-form McGill Pain Questionnaire (SF-MPQ-2) | Baseline and week 4
  The Short-form McGill Pain Questionnaire-2 is a modified version of the original SF-MPQ, assessing pain in patients with various conditions. It comprises 22 descriptors rated on a 0-10 scale, providing a comprehensive evaluation of pain. The Short Form McGill Pain Questionnaire 2 (SF-MPQ-2) has demonstrated strong internal validity.

CONTACTS AND LOCATIONS:
Overall Officials: Madhanraj Sekar, MPT, Principal Investigator — Saveetha Institute of Medical and Technical Sciences
Locations (1):
- Saveetha Institute of Medical and Technical Sciences, Chennai, Tamil Nadu, India

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT07325032/SAP_000.pdf